CLINICAL TRIAL: NCT06965127
Title: Enhancing Walking and Independence After Incomplete SCI With a Fully Implanted Neuroprosthesis
Brief Title: Implant for Walking After Incomplete SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Collaborators: MetroHealth Medical Center (Other); CDMRP (Unknown)
Responsible Party: Principal Investigator, Nathan Makowski, Associate Professor, Louis Stokes VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1802378; CDMRP-SC230198 (Other Grant/Funding Number: DoD CDMRP)
Record Dates: First submitted 2025-04-22; First posted 2025-05-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury (SCI); Gait
Keywords: neuroprosthesis; implanted device
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Implantation, controller development and evaluation (Experimental): This phase includes installing the device and setting the individual up for use of the system and evaluating the effect of the system on walking ability.
  Interventions: Device: NNP-LE

INTERVENTIONS:
Device: NNP-LE — Networked NeuroProsthesis - Lower Extremity Configuration (NNP-LE) measuring physiologic command signals and delivering neural stimulation to intramuscular and nerve cuff electrodes for trunk and leg muscle assistance.

SUMMARY:
This is a device study that will evaluate the effect of an implanted stimulator on improving walking in people with incomplete spinal cord injury. There are two phases in the study: 1) Screening - this phase determines if the individual is a good candidate to receive an implanted system, 2) Implantation, controller development, and evaluation - this phase includes implanting the device and setting the individual up for system use, creating controllers for walking, and evaluating the effect of the device over a couple years.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of neural stimulation for improving walking after incomplete spinal cord injury. Participants will conduct pre-surgical gait training and then undergo surgery to implant a stimulator and electrodes to sense from and activate muscles used during walking. The device delivers electrical pulses to the nerves causing the muscles to contract to perform functional movements. The system coordinates assistance based on implanted sensors. After receiving the implanted device, participants undergo training to use the device to assist walking. Evaluations are completed prior to surgery as well after training and at later follow up sessions.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75
* Non-ventilator dependent paralysis resulting from injuries such as: cervical/thoracic spinal cord injuries affecting the trunk and/or lower limbs
* Impairment classification of AIS B, C, or D (preservation of sensation and/or some motor function) with weakness in trunk and/or lower extremity muscles
* Unable to walk faster than 0.8m/s during a 10m walk test
* Gait deviation such as reduced peak hip, knee, and/or ankle range of motion during stance or swing phases due to motor impairment
* Time post injury greater than six months
* Innervated and excitable lower extremity and trunk musculature
* Adequate social support and stability
* Willingness to comply with follow-up procedures
* Appropriate body habitus (height and weight within acceptable limits as determined by study physician)
* Neurologically stable as determined by a physician

Exclusion Criteria:

* Significant fracture risk or history of spontaneous fractures
* History of heterotopic ossification at the hip, knee, or ankle
* Non-English speaking
* Insufficient upper extremity function to use an assistive device (e.g. walker or cane)
* Females who are pregnant
* Current pressure injury that would be exacerbated by study activities
* Uncontrolled spasticity that would interfere with study activities
* Significant range of motion limitations that would compromise study activities
* History of vestibular dysfunction, balance problems, or spontaneous falls
* Disorder or condition that require MRI monitoring
* Acute and/or untreated orthopedic issues that would prevent weight bearing or exercising implanted muscles such as a dislocation or fracture
* Acute and/or chronic medical problems left untreated or not controlled that would increase risk by using stimulation such as cardiac abnormalities, immunological/pulmonary/renal/circulatory compromise
* Uncontrolled diabetes or hypertension
* Presence of a demand pacemaker, cardiac defibrillator, or neuroprosthesis system with components in the legs
* Any other medical or psychological condition that would be a contraindication

Implant eligibility criteria

• In addition to all of the above, the participant must be able to fully support their body weight in standing with an assistive device prior to implantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Difference in maximum walking distance | Immediately after the participant is fully trained to use their implanted system
  The maximum walking distance is a measure of how far the participant can walk within a single bout over an unconstrained period of time. The measure is used to assess whether endurance and walking capacity improve. The difference between walking with and without the system turned on determines if the system improves walking capacity. Users serve as their own concurrent controls.

SECONDARY OUTCOMES:
Difference in spinal cord injury - functional ambulation inventory (SCI-FAI) | Immediately after the participant is fully trained to use their implanted system
  The SCI-FAI is an observational gait assessment that assesses three areas of walking: gait parameters, assistive device use, and walking mobility. The difference between walking with and without the system turned on determines if the system improves walking ability. Users serve as their own concurrent controls with and without device assistance.
Difference in Home and community mobility | Baseline and Immediately after the participant is fully trained to use their implanted system
  A body worn step counter measures the number of steps taken daily over the course of about a month prior to implantation and then after implantation and system use. The difference between walking before and after having the system identifies if people walk more once they have the system. Users serve as their own longitudinal controls.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Makowski, PhD, Principal Investigator — MetroHealth System, Ohio
Locations (1):
- Louis Stokes Cleveland Veterans Affairs Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified assessment data will be shared via open data commons for spinal cord injury
Time Frame: data will become available after study completion
Access Criteria: de-identified data will be available to anyone with access to the ODC-SCI repository
URL: https://odc-sci.org